CLINICAL TRIAL: NCT03057041
Title: Intranasal Fentanyl for Pain Control During First-Trimester Uterine Aspiration: A Randomized Controlled Trial
Brief Title: Intranasal Fentanyl for Pain Control During First-Trimester Uterine Aspiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INF
Record Dates: First submitted 2017-02-14; First posted 2017-02-17 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Pain Uterus
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fentanyl (Experimental)
  Interventions: Drug: Fentanyl
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Fentanyl — 100 mcg of intranasal fentanyl, 50 mcg/ mL in each nostril via mucosal atomizer 15 minutes prior to procedure start
  Arms: Fentanyl
Drug: placebo — 1 mL of sterile saline in each nostril via mucosal atomizer 15 minutes prior to procedure start
  Arms: Placebo

SUMMARY:
Intranasal fentanyl has been found to be safe and effective in the reduction of pain among pediatric and adult populations. The investigators hypothesize that patients who receive 100 mcg of intranasal fentanyl for pain control before first-trimester uterine aspiration will report lower pain scores than those who receive placebo. The investigators will test this hypothesis using a randomized, double-blind, placebo-controlled trial comparing pain reported during uterine aspiration between patients who receive either intranasal fentanyl or intranasal saline prior to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Seeking office based uterine aspiration
* Gestational age at 14 weeks or less
* Age 14 years or older with parental consent to participate in this research study if 14-17 years old
* Able to read, speak, and understand English
* Ability to understand materials and consent forms

Exclusion Criteria:

* Seeking medical abortion, operating room based surgical abortion, or operating room based miscarriage management
* Gestational age greater than 14 weeks
* Age less than 14 years old
* Inability to read, speak, and understand English
* Current incarceration
* Weight less than 40kg
* Self-reported or documentation of significant cardiopulmonary disease
* Self-reported or documentation of alcohol or substance dependence or abuse
* Contraindications, relative contraindication to fentanyl use

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Pain during uterine aspiration | During uterine aspiration or immediately after uterine aspiration
  Self reported on 100 mm VAS

SECONDARY OUTCOMES:
Patient satisfaction with procedural pain control | approximately 15 minutes after procedure ends
  Self reported on 100 mm VAS
Post-procedural pain | approximately 15 minutes after procedure end
  Self reported on 100 mm VAS

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Women's Options Center, Honolulu, Hawaii
  - Planned Parenthood Columbia Willamette, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No